CLINICAL TRIAL: NCT02439060
Title: Prevention of Parastomal Hernia Following Radical Cystectomy and Ileal Conduit Using Biologic Mesh: Randomized Clinical Trial
Brief Title: PUBMIC (Prophylactic Use of Biologic Mesh in Ileal Conduit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4B-14-2; NCI-2015-00278 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4B-14-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Bladder Carcinoma; Hernia
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hernia | interventions — Alloderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (biologic mesh) (Experimental): Patients undergo placement of biologic mesh during radical cystectomy and placement of the ileal conduit.
  Interventions: Other: Acellular Cadaveric Dermal Matrix
- Arm II (no intervention) (No Intervention): Patients undergo standard of care radical cystectomy and placement of the ileal conduit.

INTERVENTIONS:
Other: Acellular Cadaveric Dermal Matrix — Undergo intraperitoneal prophylactic mesh placement
  Other Names: ACDM; AlloDerm; DermaMatrix
  Arms: Arm I (biologic mesh)

SUMMARY:
This randomized phase III trial studies how well biologic mesh works in preventing parastomal hernia in patients with bladder cancer who are undergoing radical cystectomy, or removal of the bladder, and ileal conduit diversion. An ileal conduit is a tube created from your small intestine that will be used as a tube for urine to flow out of your body. Parastomal hernia is a type of hernia that can occur in the stomach area where the ileal conduit is placed. Biologic mesh may help prevent parastomal hernia following surgery and ileal conduit diversion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of developing parastomal hernia detected either clinically or radiologically in patients with radical cystectomy and ileal conduit, with or without mesh.

SECONDARY OBJECTIVES:

I. To estimate the rate of developing symptomatic parastomal hernia requiring surgical intervention in patients with radical cystectomy and ileal conduit with or without mesh.

II. To estimate the time from cystectomy with an ileal conduit to diagnosis of clinical parastomal hernia development in patients with radical cystectomy and ileal conduit with or without mesh.

III. To estimate the time from cystectomy with an ileal conduit to diagnosis of radiological parastomal hernia development in patients with radical cystectomy and ileal conduit with or without mesh.

IV. To estimate the rate of stomal prolapse and time to its development in patients with radical cystectomy and ileal conduit with or without mesh.

V. To evaluate mesh-related complications in mesh group.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo placement of biologic mesh during radical cystectomy and placement of the ileal conduit.

ARM II: Patients undergo standard of care radical cystectomy and placement of the ileal conduit.

After completion of study, patients are followed up every 2-4 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer, undergoing radical cystectomy and ileal conduit diversion
* Ability to understand and the willingness to sign a written informed consent
* Follow-up either here at University of Southern California (USC) or centers that are available to transfer the requested clinical and radiological data

Exclusion Criteria:

* Previous scar or mesh at the level of ileal conduit
* Survival less than 12 months after surgery (either predicted survival before surgery or actual survival after surgery < 12 months)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cadaveric component, i.e. Flex HD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Rate of development of a clinical or radiologic parastomal hernia | Up to 2 years
  Cumulative incidence curves (using death, local recurrence, other surgical procedures unrelated to the development of parastomal hernias as competing risks) and their associated estimates (at 2 years) and standard errors will be used. To compare the two arms, the Wald test for the estimate at two years will be used, and the log-rank test for the timing of the events will be used. All tests will be one-sided at the 0.05 level.

SECONDARY OUTCOMES:
Incidence of mesh-related complications in Mesh group (Arm I) | Up to 2 years
  All patients randomized, who undergo a radical cystectomy with an ileal conduit, will be classified according to whether or not they received the mesh implant. Observed toxicities and complications during and after surgery will be summarized by treatment received, severity, timing (time from surgery), and frequency.
Rate of development of symptomatic parastomal hernia requiring surgical intervention | Up to 2 years
  Cumulative incidence curves (using death, local recurrence, other surgical procedures unrelated to the development of parastomal hernias as competing risks) and their associated estimates (at 2 years) and standard errors will be used. To compare the two arms, the Wald test for the estimate at two years will be used, and the log-rank test for the timing of the events will be used. All tests will be one-sided at the 0.05 level.

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Djaladat, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States